CLINICAL TRIAL: NCT04136782
Title: Albumin-bound Paclitaxel Combined With Carboplatin Versus Epirubicin Combined With Docetaxel as Neoadjuvant Therapy for Triple-negative Breast Cancer: a Multicenter Randomized Controlled Phase IV Clinical Trial
Brief Title: Albumin-bound Paclitaxel and Carboplatin Versus Epirubicin and Docetaxel for Triple-negative Breast Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Principal Investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Shengjing-LCG005
Record Dates: First submitted 2019-10-22; First posted 2019-10-23 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: adjuvant chemotherapy; paclitaxel; albumin-bound paclitaxel; carboplatin; docetaxel; epirubicin
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Experimental): 55 cases of triple-negative breast cancer will be assigned into a trial group.
  Interventions: Drug: Albumin-bound paclitaxel combined with carboplatin
- Control group (Active Comparator): 55 cases of triple-negative breast cancer will be assigned into a control group.
  Interventions: Drug: Epirubicin combined with docetaxel

INTERVENTIONS:
Drug: Albumin-bound paclitaxel combined with carboplatin — Albumin-bound paclitaxel combined with carboplatin: Albumin-bound paclitaxel (Abraxis BioScience, LLC., Mclrose Park, IL, USA; certificate number: H20091059) will be intravenously administered at 125 mg/m2 for 30 minutes on days 1 and 8 of each 21-day session of treatment. There will be six 21-day sessions of treatment. At the same time, carboplatin (Qilu Pharmaceutical Co., Ltd., Jinan, Shandong Province, China; National Drug Approval Number: H20020181) will be intravenously administered at AUC = 2 mg•min/mL for 120 minutes on days 1 and 8 of each 21-day session of treatment. Carboplatin must be hydrated for 3 days before use to prevent nephrotoxicity.
  Other Names: Albumin-bound paclitaxel+carboplatin group
  Arms: Trial group
Drug: Epirubicin combined with docetaxel — Epirubicin (Pfizer Pharmaceutical (Wuxi) Co., Ltd., China; National Drug Approval Number: H20000496) will be intravenously administered at 90 mg/m2 for 120 minutes on day 1 of each 21-day session of treatment. At the same time, docetaxel (Sanofi-aventis Deutschland GmbH, Frankfurt am Main, Germany; National Drug Approval Number: J20150083) will be intravenously administered at 75 mg/m2 for 120 minutes. Drug administration will be performed once every other 3 weeks for four times.
  Other Names: Epirubicin+docetaxel group
  Arms: Control group

SUMMARY:
To investigate the efficacy of albumin-bound paclitaxel combined with carboplatin versus epirubicin combined with docetaxel as neoadjuvant therapy for triple-negative breast cancer.

DETAILED DESCRIPTION:
Triple-negative breast cancer is named because of lack of expression of estrogen receptor, progesterone receptor, and proto-oncogene HER2. This type of breast cancer is highly heterogeneous, is more likely to recur locally and develop distant metastasis, and has high invasiveness and low survival rate. Because both endocrine therapy and targeted therapy are ineffective for triple-negative breast cancer, so the main currently available treatment is chemotherapy. Some patients may choose anti-angiogenic therapy. The prognosis of triple-negative breast cancer is worse than that of other types of breast cancer due to fewer treatment options. Guidelines and Specifications for Diagnosis and Treatment of Breast Cancer (2017 edition) compiled by Committee of Breast Cancer Society of Chinese Anti-Cancer Association suggest that neoadjuvant therapy should be recommended for patients with large-sized tumors (maximum diameter greater than 5 cm), axillary lymph node metastasis, human epidermal growth factor receptor 2 (HER-2) positive, triple-negative breast cancer, and breast-conserving intention. The guidelines also suggest that neoadjuvant therapy for triple-negative breast cancer should apply anthracyclines and taxanes. Guidelines of Chinese Society of Clinical Oncology (CSCO) Breast Cancer 2018.V1 propose that the treatment regimen of triple-negative breast cancer should apply anthracyclines and taxanes. The treatment regimens of taxanes, anthracyclines, and cyclophosphamides in combination (1A) or taxanes combined with anthracyclines (2A) are strongly recommended. In 2015, St Gallen recommended anthracyclines and taxanes as the main chemotherapeutic drugs for triple-negative breast cancer. However, the pathologic complete remission (pCR) rate of paclitaxel combined with anthracycline as neoadjuvant therapy was still less than 50%. In the GALGB40603 study, the pCR rate of breast and axillary lymph nodes increased from 41% to 54% with carboplatin based on standard chemotherapeutic drugs anthracycline combined with taxanes. The Gepar Sixto-GBG 66 study also suggested that carboplatin could increase the pCR rate in triple-negative breast cancer patients. Compared with other dosage forms of paclitaxel, albumin-bound paclitaxel can produce higher paclitaxel concentration in local tumors, and the injection time is shorter. At present, the drug has been approved by the Food and Drug Administration of the United States for adjuvant chemotherapy for breast cancer with metastasis or recurrence within 6 months that fails to respond to combined chemotherapy. However, little is currently reported on albumin-bound paclitaxel combined with carboplatin versus anthracycline combined with paclitaxel in China. A multicenter randomized controlled phase IV clinical trial will be conducted to investigate the efficacy of albumin-bound paclitaxel combined with carboplatin versus epirubicin combined with docetaxel as neoadjuvant therapy for triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients developing breast cancer as confirmed by X-ray examination, cancer tissue negative for estrogen receptor, progesterone receptor and HER2, and tumor stage II-III;
* estimated survival > 3 months;
* presence of clinically measurable lesions;
* Karnofsky functional status score ≥ 70;
* normal routine blood test results, normal liver and kidney function, and near normal electrocardiographic manifestations;
* age at 18-70 years.

Exclusion Criteria:

* stage IV breast cancer patients with bone metastasis or other distant metastasis;
* severe renal insufficiency;
* older adult patients with severe organic diseases such as heart and lung diseases, who are not estimated to be able to tolerate chemotherapy;
* those who have received antineoplastic therapy;
* those who have received neoadjuvant chemotherapy but fail in 2 cycles of neoadjuvant chemotherapy and switch to other regimens or terminate chemotherapy;
* those with history of other malignant tumors;
* those with severe heart, liver, and kidney organ dysfunction or poor health who cannot tolerate chemotherapy, or those who cannot tolerate chemotherapy and switch to other therapeutic regimens;
* those with mental and nervous system diseases who cannot comply with treatment;
* those with dexamethasone intolerance or those who are highly allergic to any drug in neoadjuvant chemotherapy;
* pregnant or lactating women;
* those who are participating in other trials.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Estimated)
Dates: Start 2021-07-19 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete remission rate | 5 years after treatment
  Pathologic complete remission will be evaluated 5 years after treatment according to the regression of tumors. Tumor regression will be assessed according to RECIST 1.1. Complete remission (CR)

SECONDARY OUTCOMES:
Breast-conserving rate | After 6 months of treatment
  The percentage of patients with breast conservation after 6 months of treatment.
Incidence of osteoporosis | Every 6 months for 5 successive years
  Osteoporosis is considered to be present when a patient's bone density or bone mineral content is more than 2.5 standard deviations below the mean value of normal adult bone density. Patients will be screened for osteoporosis once every 6 months for 5 successive years. Incidence of osteoporosis = number of patients developing osteoporosis/total number of patients ×100%
Incidence of bone-related events | Every 6 months for 5 successive years
  Bone pain, fracture and other bone related events. Patients will be screened for bone-related events once every 6 months for 5 successive years. Incidence of bone-related events = number of patients having bone-related events/total number of patients × 100%.
Incidence of other distant organ metastasis related events | Every 6 months for 5 successive years
  Metastasis to other distant organs such as the lung, liver, bone marrow, brain, and ovary. Patients will be screened for other distant organ metastasis related events once every 6 months for 5 successive years. Incidence of other distant organ metastasis related events = number of patients having other distant organ metastasis related events/total number of patients × 100%.
Disease-free survival (DFS) | Within 5 years after disease onset.
  The time from the start of the enrollment to the recurrence of the disease or the death of the patient due to disease progression. DFS will be analyzed according to the specific situation within 5 years after disease onset.
Overall survival (OS) | Within 5 years after disease onset.
  The time from the start of the enrollment to the death of the patient: OS will be analyzed according to the specific situation within 5 years after disease onset.
Adverse events | in 5 years
  Any untoward medical occurrence in a patient and which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Caigang Liu, M.D., Ph.D., Principal Investigator — Shengjing Hospital
Locations (7):
- China (7):
  - Cancer Hospital Affiliated to Harbin Medical University, Harbin, Heilongjiang
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - Panjin Liaohe Oilfield Gem Flower Hospital, Panjin, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning